CLINICAL TRIAL: NCT00241839
Title: Uric Acid and Hypertension in African Americans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 332; R01HL079352 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Allopurinol; Sugars; Chlorthalidone; Potassium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Chlorthalidone 25 mg and Potassium Chloride 40-50meq were given daily for 5 weeks before baseline visit for testing. After baseline testing was completed, Allopurinol 300mg daily was added for 8-10 weeks at which time testing was repeated.
  Interventions: Drug: Allopurinol; Drug: Chlorthalidone; Drug: Potassium chloride
- B (Placebo Comparator): Chlorthalidone 25 mg and Potassium Chloride 40-50meq were given daily for 5 weeks before baseline visit for testing. After baseline testing was completed, a Placebo,matched in appearance to Allopurinol, was added daily for 8-10 weeks, at which time testing was repeated.
  Interventions: Drug: Placebo; Drug: Chlorthalidone; Drug: Potassium chloride

INTERVENTIONS:
Drug: Allopurinol — Allopurinol (300 mg capsule) was given for 8-10 weeks compared to placebo group after initial baseline testing. After two weeks on the Allopurinol, a serum uric acid level was obtained. If the uric acid level was greater than 5.5, the Allopurinol dosage was increased to 600mg (two 300 mg capsules)for the duration of the trial, 6-8 weeks.
  Other Names: Zyloprim
  Arms: A
Drug: Placebo — Placebo capsule (matched in appearance for Allopurinol and labeled 300mg) was given for 8-10 weeks compared to the Allopurinol group after initial baseline testing. After two weeks on the placebo, a serum uric acid level was obtained. If the uric acid level was greater than 5.5, the placebo dosage was increased to 600mg (two 300 mg capsules)for the duration of the study, 6-8 weeks.
  Other Names: sugar pill
  Arms: B
Drug: Chlorthalidone — Chlorthalidone 25 mg was given daily for 5 weeks before baseline visit for testing and continued through out the study.
Drug: Potassium chloride — Potassium Chloride 40-50meq was given daily for 5 weeks before baseline visit for testing and continued through out the study.

SUMMARY:
This study will test the hypothesis that the administration of a xanthine oxidase inhibitor (allopurinol) will prevent thiazide-induced hyperuricemia, which will result in better blood pressure (BP) control in African Americans.

DETAILED DESCRIPTION:
Thiazide diuretics when used in the treatment of hypertension are associated with many metabolic side effects, including hyperuricemia, gout, insulin resistance, and hyperlipidemia. Each of these conditions is already highly prevalent in African Americans. Our hypothesis is that thiazide-induced hyperuricemia decreases the efficacy of thiazides in controlling BP, leads to endothelial dysfunction, and increases the incidence of insulin resistance and impaired glucose tolerance. This hypothesis will be tested in a randomized, double-blind, placebo-controlled clinical trial of 8-10 weeks duration in which a total of 100 African American patients with hypertension will be enrolled, randomized, and treated as follows:

1. Subjects with untreated stage I hypertension will receive chlorthalidone (25 mg/day) and potassium chloride (40 mEq/day) for 4 weeks. Serum potassium levels will be obtained after four weeks on chlorthalidone. If the level is below 3.5 mEg/L, a bolus of 40 mEq potassium 2 to 3 times daily will be given for 2 to 3 days, or as clinically indicated. A maintenance dose of 50 mEq will be initiated. After at least 7 days, they will then be randomized to add-on allopurinol (300 mg/day) or placebo. Treatment will continue for 8-10 weeks with the chlorthalidone, potassium chloride, and allopurinol/placebo regimen.
2. Subjects with hypertension controlled (i.e. BP <140/90) or no higher than stage 1 hypertension (i.e., <160/100) on a single antihypertensive agent or two antihypertensive agents will be switched from their prior antihypertensive agent to chlorthalidone 25 mg/day, and potassium chloride (40mEq/day) for 4 weeks. Serum potassium levels will be obtained after four weeks on chlorthalidone. If the level is below 3.5 mEg/L, a bolus of 40 mEq potassium 2 to 3 times daily will be given for 2 to 3 days, or as clinically indicated. A maintenance dose of 50 mEq will be initiated. After at least 7 days, they will then be randomized to add-on allopurinol (300 mg/day) or placebo. Treatment will continue for 8-10 weeks with the chlorthalidone, potassium chloride, and allopurinol/placebo regimen.

The allopurinol (or placebo) dose will be adjusted to achieve serum uric acid levels between 4 and 5.5 mg/dL after 2 weeks on drug. All subjects will receive a low-sodium diet. The primary endpoint is reduction in systolic BP. Secondary endpoints measure endothelial function, ambulatory blood pressure, body composition, systemic inflammation, metabolic parameters, oxidant stress, and renal hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* African American (including black individuals born in the Caribbean, Africa, Canada, etc.)
* Are either untreated with any antihypertensive agent, with an average sitting clinic BP of between 140/90 and 159/99 mm Hg OR subjects with hypertension controlled (i.e. BP less than 140/90) or no higher than stage 1 hypertension (i.e., less than 160/100) on a single antihypertensive agent or two antihypertensive agents (individuals on fixed dose ARB-diuretic or ACEI-diuretic combinations will also be considered as being on monotherapy for purposes of the study. Individuals on beta blockade or calcium channel blockade for coronary artery disease and/or arrhythmia will not be eligible for the study)
* Random spot urine protein/creatinine ratio of less than 0.5 (approximates a 24-hour urinary protein excretion of 500 mg/day)
* Calculated MDRD GFR of greater than or equal to 60 ml/min/1.73/m^2
* No allopurinol or probenecid intake for at least one month prior to study entry
* Willing and able to cooperate with study procedures
* Willing to travel to the GCRC at Shands Hospital for overnight inpatient stays on two separate occasions

Exclusion Criteria:

* History of malignant or accelerated hypertension
* Confirmed total white cell count of less than 2,500/mm^3, anemia, or thrombocytopenia
* Known history of liver disease
* Known secondary cause of hypertension
* Known presence of diabetes or fasting blood glucose greater than or equal to 126 mg/dL
* History of heart failure, acute myocardial infarction, or stroke or on a β-blocker or calcium channel blocker for cardiovascular indications other than for lowering blood pressure
* Abnormal EKG requiring medical intervention
* History of clinical or renal biopsy or evidence of renal parenchymal disease
* Acute gout attack within 2 weeks of study entry
* History of drug abuse in the last 2 years, including narcotics, cocaine, or alcohol (greater than 21 drinks/week)
* Arm circumference of greater than 52 cm, which precludes measurement with a 'thigh' BP cuff
* History of a reaction to allopurinol or chlorthalidone
* Pregnant or planning to become pregnant during the study, or breastfeeding
* History of noncompliance, are unable to comply with the study requirements, or who are currently participating in another study
* Not fasting prior to obtaining screening laboratory data. If a participant has clearly not fasted, we will exclude those individuals with casual blood glucose levels of greater than or equal to 200 mg/dL. In the event that a fasting blood sugar exceeds 126 mg/dL, it will be reconfirmed on a blood glucose measurement obtained on a subsequent day, per American Diabetes Association criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Segal, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Johnson RJ, Segal MS, Sautin Y, Nakagawa T, Feig DI, Kang DH, Gersch MS, Benner S, Sanchez-Lozada LG. Potential role of sugar (fructose) in the epidemic of hypertension, obesity and the metabolic syndrome, diabetes, kidney disease, and cardiovascular disease. Am J Clin Nutr. 2007 Oct;86(4):899-906. doi: 10.1093/ajcn/86.4.899. PMID 17921363
- [Background] Nakagawa T, Johnson RJ. Hypertension: Is there a dark side to thiazide therapy for hypertension? Nat Rev Nephrol. 2010 Oct;6(10):564-6. doi: 10.1038/nrneph.2010.114. No abstract available. PMID 20871636
- [Background] Nakagawa T, Kang DH, Feig D, Sanchez-Lozada LG, Srinivas TR, Sautin Y, Ejaz AA, Segal M, Johnson RJ. Unearthing uric acid: an ancient factor with recently found significance in renal and cardiovascular disease. Kidney Int. 2006 May;69(10):1722-5. doi: 10.1038/sj.ki.5000391. PMID 16598194
- [Background] Reungjui S, Hu H, Mu W, Roncal CA, Croker BP, Patel JM, Nakagawa T, Srinivas T, Byer K, Simoni J, Wesson D, Sitprija V, Johnson RJ. Thiazide-induced subtle renal injury not observed in states of equivalent hypokalemia. Kidney Int. 2007 Dec;72(12):1483-92. doi: 10.1038/sj.ki.5002564. Epub 2007 Oct 10. PMID 17928827
- [Background] Reungjui S, Roncal CA, Mu W, Srinivas TR, Sirivongs D, Johnson RJ, Nakagawa T. Thiazide diuretics exacerbate fructose-induced metabolic syndrome. J Am Soc Nephrol. 2007 Oct;18(10):2724-31. doi: 10.1681/ASN.2007040416. Epub 2007 Sep 12. PMID 17855639
- [Background] Kim KM, Henderson GN, Frye RF, Galloway CD, Brown NJ, Segal MS, Imaram W, Angerhofer A, Johnson RJ. Simultaneous determination of uric acid metabolites allantoin, 6-aminouracil, and triuret in human urine using liquid chromatography-mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Jan 1;877(1-2):65-70. doi: 10.1016/j.jchromb.2008.11.029. Epub 2008 Nov 25. PMID 19081307
- [Background] Kim KM, Henderson GN, Ouyang X, Frye RF, Sautin YY, Feig DI, Johnson RJ. A sensitive and specific liquid chromatography-tandem mass spectrometry method for the determination of intracellular and extracellular uric acid. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Jul 15;877(22):2032-8. doi: 10.1016/j.jchromb.2009.05.037. Epub 2009 May 27. PMID 19520625
- [Derived] Fravel MA, Ernst ME. Management of gout in the older adult. Am J Geriatr Pharmacother. 2011 Oct;9(5):271-85. doi: 10.1016/j.amjopharm.2011.07.004. Epub 2011 Aug 17. PMID 21849262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was through flyers and voluntary blood pressure checks and hypertension lectures throughout the county in churches, health fairs, community art festivals, new business openings and celebrations, and in hospital lobbies, business employee lounges, store front spaces at grocery stores and super stores. Individuals also self-refered.
Pre-assignment Details: 150 subjects signed consents;8 were withdrawn prior to randomization. All participants were placed on chlorthalidone 25mg daily for blood pressure stabilization along with potassium chloride (KCL) 40meq daily. Potassium chloride was increased to 50meq daily for those subjects whose serum potassium was less than 3.5 before baseline visit.
Groups:
- A (Allopurinol): Chlorthalidone 25 mg and Potassium Chloride 40-50meq were given daily for 5 weeks before baseline visit for testing. After baseline testing was completed, Allopurinol 300mg daily was added for 8-10 weeks. Serum uric acid (UA) levels were checked at study visit 2 weeks post baseline. If UA levels were above 5.0 an additional 300mg allopurinol was added with total dose of 600mg daily. The dosage of allopurinol then remained constant throughout the remainder of the study. Testing was repeated at 8-10 weeks after baseline.
- B(Placebo): Chlorthalidone 25 mg and Potassium Chloride 40-50meq were given daily for 5 weeks before baseline visit for testing. After baseline testing was completed, a Placebo, having the same appearance and dosage label(300mg)as allopurinol, was added for 8-10 weeks. Serum uric acid (UA) levels were checked at study visit 2 weeks post baseline. If UA levels were above 5.0 an additional placebo (300mg)was added with total dose of 600mg daily. The dosage of placebo then remained constant throughout the remainder of the study. Testing was repeated at 8-10 weeks after baseline.
Period: Overall Study
Arm/Group | A (Allopurinol) | B(Placebo)
Started | 71 | 71
Completed | 52 (N=52 represents number with both baseline and 8-10 week data. N<52 implies missing data.) | 53 (N=53 represents number with both baseline and 8-10 week data. N<53 implies missing data.)
Not Completed | 19 | 18
Not completed — Withdrawal by Subject | 18 | 17
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: African Americans with borderline high Blood Pressure
Groups:
- B (Placebo): Chlorthalidone 25 mg and Potassium Chloride 40-50meq were given daily for 5 weeks before baseline visit for testing. After baseline testing was completed, a Placebo, having the same appearance and dosage label(300mg)as allopurinol, was added for 8-10 weeks. Serum uric acid (UA) levels were checked at study visit 2 weeks post baseline. If UA levels were above 5.0 an additional placebo (300mg)was added with total dose of 600mg daily. The dosage of placebo then remained constant throughout the remainder of the study. Testing was repeated at 8-10 weeks after baseline.
- Total: Total of all reporting groups
Arm/Group | A (Allopurinol) | B (Placebo) | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 71 | 141
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.1) | 48.0 (7.7) | 47.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  United States | 71 | 71 | 142

OUTCOME MEASURES:

1. Primary Outcome: Change in Diastolic Blood Pressure by Cuff 8-10 Weeks Minus Baseline
Description: The Diastolic BP was taken at Baseline and after 8-10 weeks of treatment or placebo while on chlorthalidone and potassium chloride. The blood pressure was measured according to "Shared Care" protocol: 15 minutes of quiet, undisturbed rest with three BP measurements obtained subsequently at 5 minute intervals.
  The mean of the second and third reading was the value used for analysis for both the Baseline measurement and the measurement after 8 - 10 weeks of treatment. The dependent variable is baseline value minus ending value.
  Measures are in millimeters of mercury (mm hg)
Time Frame: Measured at 8-10 weeks on allopurinol / placebo
Population: Participants were individuals with essential hypertension (BP 140/90-160/100) on none or up 2 antihypertensive drugs without any other chronic condition or illness. For their data to be included in analysis they had to complete the study (includes baseline to last visit).
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- B (Placebo): Chlorthalidone 25 mg and Potassium Chloride 40-50meq were given daily for 5 weeks before baseline visit for testing. After baseline testing was completed, Placebo 300mg daily (identical in size, color, and dosage as allopurinol) was added for 8-10 weeks. Serum uric acid (UA) levels were checked at study visit 2 weeks post baseline. If UA levels were above 5.0 an additional 300mg placebo was added with total dose of 600mg daily. The dosage of placebo then remained constant throughout the remainder of the study. Testing was repeated at 8-10 weeks after baseline.
Arm/Group | A (Allopurinol) | B (Placebo)
Number analyzed (Participants) | 52 | 53
mm Hg | 3.44 (12.25) | -0.83 (10.63)
Statistical Analysis 1: Comparison: A (Allopurinol) vs B (Placebo); We compared the drop in baseline of diastolic BP for the two treatment groups Allopurinol vs. Placebo by a Satterthwaite corrected t-test; Test type: Superiority or Other; p = 0.059, t-test, 2 sided; Satterthwaite correction for possibly unequal variance was made; Mean Difference (Net) = 4.27, 95% CI 2-sided [-0.17 to 8.7], Standard Error of Mean 2.24 — A positive value of the estimated value would favor the allopurinol arm. The analysis is limited to those with both baseline and 8-10 week data on this variable

2. Primary Outcome: Change in Systolic Blood Pressure by Cuff After 8-10 Weeks Minus Baseline
Description: The systolic BP was taken at Baseline and after 8-10 weeks of treatment on placebo, while on chlorthalidone and potassium chloride. The blood pressure was measured according to "Shared Care" protocol: 15 minutes of quiet, undisturbed rest with three BP measurements obtained subsequently at 5 minute intervals.
  The mean of the second and third reading was the value used for analysis for both the Baseline measurement and the measurement after 8 - 10 weeks of treatment. The dependent variable is baseline value minus ending value.
  Measures are in millimeters of mercury (mm hg)
Time Frame: Measured at 8-10 weeks on allopurinol or placebo
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | A (Allopurinol) | B (Placebo)
Number analyzed (Participants) | 52 | 53
mm Hg | 0.21 (7.37) | -0.95 (8.90)
Statistical Analysis 1: Comparison: A (Allopurinol) vs B (Placebo); Test type: Superiority or Other; p = 0.47, t-test, 2 sided — Positive numbers indicate a drop. We compared baseline minus value at treatment end for the two treatments; Satterthwaite correction was used for potentially unequal variances; Mean Difference (Net) = 1.16, 95% CI 2-sided [-2.0 to 4.3], Standard Error of Mean 1.59 — The analysis is limited to those with both baseline and 8-10 week data on this variable

3. Secondary Outcome: Change in Overall Mean BP From Those Obtained by 24 Hour Ambulatory Blood Pressure Measurements (ABPM) 8-10 Weeks Minus Baseline.
Description: Subjects had 24 hr blood pressure monitoring (ABPM) at baseline and treatment end. The readings were averaged and the changes from baseline to treatment end were compared.
Time Frame: Baseline and end of treatment (8-10 weeks on allopurinol / placebo)
Population: We obtained over 90% of those with cuff measures on the 24 hour BP measures (ABPM).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | A (Allopurinol) | B (Placebo)
Number analyzed (Participants) | 49 | 50
mm Hg | -5.9 (11.9) | 0.90 (8.91)
Statistical Analysis 1: Comparison: A (Allopurinol) vs B (Placebo); Test type: Superiority or Other; p = 0.0020, t-test, 2 sided; Sattherthwaite correction was used; Median Difference (Net) = -6.76, 95% CI 2-sided [-11.0 to -2.6], Standard Error of Mean 2.11 — The analysis is limited to those with both baseline and 8-10 week data on this variable. The 24 hour was in the opposite direction of the cuff

4. Secondary Outcome: Change in Uric Acid (UA) Levels: Baseline Less End of Treatment
Description: Subjects on allopurinol are expected to lower their uric acid levels relative to placebo.
Time Frame: Baseline UA levels compared to end of treatment levels (8-10 weeks on allopurinol / placebo)
Population: Change in uric acid from baseline to end of treatment.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | A (Allopurinol) | B (Placebo)
Number analyzed (Participants) | 50 | 53
mg/dl | 2.29 (1.29) | 0.14 (0.88)
Statistical Analysis 1: Comparison: A (Allopurinol) vs B (Placebo); We expected allopurinol to be associated with a decrease in uric acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Satterthwaite correction was used; Median Difference (Net) = 2.15, 95% CI 2-sided [1.72 to 2.59], Standard Error of Mean 0.22 — Allopurinol was associated with a significant decrease in uric acid over the treatment period as compared to placebo. The analysis is limited to those with both baseline and 8-10 week data on this variable

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 5 years, 1 month which represents the time the first consent was signed until the last subject completed participation in the study.
Arm/Group | A (Allopurinol) | B (Placebo)
Serious Adverse Events (participants affected / at risk) | 4/71 | 3/71
Other Adverse Events (participants affected / at risk) | 26/71 | 11/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (Allopurinol) (N=71) | B (Placebo) (N=71)
Fatigue (Nervous system disorders) | 0 (0) | 1 (1)
Panic Attack (Nervous system disorders) | 1 (1) | 0 (0) — Occurred before treatments diverged.
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) — Occurred before treatments diverged.
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Occurred before treatments diverged.
Car Accident (Social circumstances) | 1 (1) | 0 (0) — Occurred before treatments diverged. Was passenger
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — Subject was hospitalized after feeling dizzy, nauseous, sweating and fainting. He regained consciousness after 1-2 minutes. All workups at the hospital were negative. After fluid hydration, he returned to his usual state of health.
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject experienced a rash beginning on her arms and chest throughout her body in her last week of treatment in the study. The dermatologist diagnosed drug reaction, but could not determine which of several drugs, including study drugs, it was.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (Allopurinol) (N=71) | B (Placebo) (N=71)
Headache (General disorders) | 7 (7) | 6 (6)
Musculoskeletal pain/ache (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (3)
Cold (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3)

LIMITATIONS AND CAVEATS:
For all 4 outcomes analyzed, patients required to have data at both baseline and 8-10 weeks on that field to be included. Thus, the numbers of subjects varies slightly from analysis to analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No